CLINICAL TRIAL: NCT03125460
Title: Clinical Evaluation of Xpert Bladder Cancer Monitor for Monitoring the Recurrence of Bladder Cancer
Brief Title: Clinical Evaluation of a Test for Monitoring the Recurrence of Bladder Cancer
Status: Completed | Type: Observational
Sponsor: Cepheid (Industry)
Responsible Party: Sponsor
Other Study IDs: 170
Record Dates: First submitted 2017-04-17; First posted 2017-04-24 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Initial Enrollment: Initial enrollment of patients with history of bladder cancer
  Interventions: Device: Xpert Bladder Cancer Monitor
- Longitudinal Cohort: Longitudinal Cohort - patients considered anticipatory positive at the time of enrollment and one random disease negative patient per anticipatory positive patient
  Interventions: Device: Xpert Bladder Cancer Monitor

INTERVENTIONS:
Device: Xpert Bladder Cancer Monitor — in vitro diagnostic test for the recurrence of bladder cancer in patients that have been previously diagnosed with bladder cancer

SUMMARY:
The objective of this study is to establish the performance characteristics of an assay that detects the recurrence of bladder cancer in patients previously diagnosed with bladder cancer. The study is conducted at locations within and outside of the United States. Testing is performed on urine specimens provided by eligible enrolled patients. Results from this study will not be used for patient management decisions.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 40 years of age
* Subject has provided documented informed consent as required by the reviewing IRB or EC. Experimental Bill of Rights will be documented for all subjects enrolled in applicable states.
* Subject is considered disease positive within 12 months (365 days) of enrollment.
* At the time of the enrollment visit, the subject is scheduled for a standard of care cystoscopy which will be completed within 3 days of providing a urine specimen.
* Subject has agreed to provide at least 60 mL of voided urine for study purposes at the enrollment visit.
* Subject has agreed to provide at least 60 mL of voided urine for study purposes at each subsequent standard of care cystoscopy visit for at least 12 months (365 days) following enrollment if the subject will enter the Longitudinal cohort.
* Any subject considered anticipatory positive at the initial visit shall be enrolled into the longitudinal cohort. For each anticipatory positive enrolled into the longitudinal cohort a random disease negative subject shall be enrolled.

Exclusion

* Subject has been previously enrolled into the study.
* Urine specimen to be used for study purposes is from the first morning void.
* Subject has had an excision procedure within six weeks (42 days) of enrollment.
* The subject is not scheduled for a standard of care cystoscopy visit within 12 months (365 days) following enrollment.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Urology clinics
Sampling Method: Non-Probability Sample
Enrollment: 424 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Comparison to histology for positive or suspicious cystoscopy | Baseline = Subject Enrollment
  Comparison to histology for positive or suspicious cystoscopy
Comparison to histology for positive or suspicious cystoscopy | Follow up = 12 months from Subject Enrollment (Baseline)
  Comparison to histology for positive or suspicious cystoscopy

SECONDARY OUTCOMES:
Comparison to UroVysion and urine cytology | Baseline = Subject Enrollment
  Urovysion and urine cytology
Comparison to UroVysion and urine cytology | Follow up = 12 months from Subject Enrollment (Baseline)
  Urovysion and urine cytology

CONTACTS AND LOCATIONS:
Locations (17):
- United States (11):
  - PAVA, Palo Alto, California
  - The Urology Center of Colorado, P.C., Denver, Colorado
  - Urology Associates, P.C., Englewood, Colorado
  - North Idaho Urology, Coeur d'Alene, Idaho
  - Idaho Urologic Institute, Meridian, Idaho
  - UroPartners, Melrose Park, Illinois
  - Five Valleys Urology, Missoula, Montana
  - Weill Cornell Medicine, New York, New York
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - UT Southwestern, Dallas, Texas
  - Virginia Urology, Richmond, Virginia
- Canada (5):
  - The Male/Female Health and Research Centre, Barrie, Ontario
  - G Kenneth Jansz Medicine Professional Corp., Burlington, Ontario
  - Urology Associates / Urologic Medical Research, Kitchener, Ontario
  - Urology Clinic of Dr. Goldfarb, North Bay, Ontario
  - Urologic Clinic of Stanley Flax, North York, Ontario
- Radboud University Medical Center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No